CLINICAL TRIAL: NCT00006471
Title: A Phase II Study of Fenretinide in Recurrent and Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Fenretinide in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-334; U01CA070172 (NIH); P30CA016672 (NIH); MDA-ID-99334 (Other: UT MD Anderson Cancer Center); NCI-610; CDR0000068294 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-11-06; First posted 2003-01-27 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Cancer
Keywords: untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the nasopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fenretinide (Experimental)
  Interventions: Drug: Fenretinide

INTERVENTIONS:
Drug: Fenretinide — 1800 mg/m2 per day for seven consecutive days, in two divided doses of 900 mg/m2 12 hours apart, repeated every 3 weeks.
  Other Names: 4-HPR

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of fenretinide in treating patients who have recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate, time to progression, median survival, and percent of 1-year survival in patients with recurrent or metastatic squamous cell carcinoma of the head and neck treated with fenretinide.
* Determine the pharmacokinetics and safety of this drug in these patients.

OUTLINE: Patients receive oral fenretinide every 12 hours on days 1-7. Treatment repeats every 3 weeks for at least 3 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response continue treatment for 1 year.

PROJECTED ACCRUAL: A total of 16-35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven recurrent squamous cell carcinoma of the head and neck
2. Stage 4 disease, either at initial presentation or at recurrence. Patients with metastatic disease at initial presentation must have received at least one prior course of cytotoxic chemotherapy.
3. Patients who present with metastatic disease should have received no more than one prior regimen of chemotherapy or biologic therapy to be eligible. Patients who initially received adjuvant or induction chemotherapy and then recurred may have received one additional cycle of chemotherapy or biologic therapy at the time of recurrence. Patients may have received any number of cycles of a particular regimen of chemotherapy.
4. Patients must have a life expectancy of at least 3 months
5. Biopsy of the recurrent lesion(s) is encouraged but not mandatory for enrollment.
6. Performance status grade 0-2.
7. Serum creatinine <= 1.5 mg/dL.
8. Serum transaminases and bilirubin <= 1.5 time normal.
9. Age >= 18 years.
10. White blood cell count >= 3,000; platelets >= 100,000; hemoglobin >= 9mg/dl.
11. Signed informed consent.
12. Women of childbearing potential must agree to utilize two methods of effective birth control, one barrier, one hormonal, or should abstain from sexual intercourse that could result in pregnancy. Contraceptive measures should be continued for at least one month after fenretinide administration has been discontinued.
13. It is recommended that male patients with female partners of childbearing potential use barrier contraception while on fenretinide.

Exclusion Criteria:

1. Pregnant women (women of childbearing potential must have a negative pregnancy test within 24 hours prior to enrollment in the study); women who are currently breast-feeding.
2. Grade 2 or greater peripheral neuropathy
3. Concurrent treatment with cytotoxic chemotherapy or radiation
4. Serious infection or other intercurrent illness requiring immediate therapy.
5. Inability to take oral medications, or other medical or social factors interfering with compliance.
6. Patients on high dose synthetic or natural Vitamin A derivatives (>= 10,000 per day).
7. Patients should not take any anti-oxidants such as Vitamin C or E.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2000-09; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To determine the response rate, time to progression, median survival, and percent one-year survival | one-year survival
  To determine the response rate, time to progression, median survival, and percent one-year survival.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org